CLINICAL TRIAL: NCT01225354
Title: An Open-label, Prospective, Postmarket Study to Assess Altering First Impressions and Self-esteem Following Radiesse® Injections.
Brief Title: Injectable Filler for Cheek Flattening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DeNova Research (Other)
Collaborators: Merz Aesthetics Inc. (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Medical Director, DeNova Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD-IMP-001
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Malar Deficiency
Keywords: Cheek; Cheek flattening; Malar deficiency; Filler
MeSH Terms: interventions — Durapatite; Prolaryn Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium hydroxylapatite (Experimental): Subject will be treated at baseline and, if needed, at 2 weeks.
  Interventions: Drug: Calcium hydroxylapatite

INTERVENTIONS:
Drug: Calcium hydroxylapatite — Subjects will be treated to full correction at visit 1 and, if needed, a touch-up injection at 2 weeks.
  Other Names: Radiesse; CaHA

SUMMARY:
The purpose of this study is to determine if Radiesse injections to the cheeks result in an altered and improved first impression and self esteem.

ELIGIBILITY:
Inclusion Criteria:

* Females between 30 and 65 years of age with Fitzpatrick Skin Color Types (I-VI).
* Have bilateral, fully visible aging defects in the malar area, corresponding to a rating of moderate to severe on the SOBER scale.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1 and be willing able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following is documented on the medical history:
* postmenopausal for at least 12 months prior to study drug administration
* without a uterus and/or both ovaries
* has had a bilateral tubal ligation for at least 6 months prior to study drug administration.
* absence of an other physical condition according to the PI's discretion
* Willingness and ability to provide written photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

* Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
* Subjects with a known allergy or sensitivity to any component of the study medications or anesthesia.
* Subjects who have had prior exposure to any calcium hydroxylapatite, or any other filler, injection for any purpose in the 12 months preceding study enrollment through the duration of the study (excluding study drug).
* Subjects who have had a prior cosmetic procedure to improve malar eminence deficiency (i.e., rhytidectomy, lower eyelid surgery, cheek implants, CO2/erbium laser resurfacing, Thermage/Thermacool radiofrequency treatment) or who have visible scars that may affect evaluation of response and/or quality of photography.
* Subjects who have had soft tissue augmentation of the malar area in the previous 6 months.
* Permanent or semi-permanent dermal fillers in the malar area.
* Ablative skin resurfacing on the malar area within the previous 6 months or during the study.
* Retinoid, microdermabrasion, or prescription level glycolic acid treatments to the malar area within 2 weeks prior to study participation or during the study.
* Active infection in the malar area (e.g., acute acne lesions or ulcers).
* Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
* Current history of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the Investigator's opinion, have a history of poor cooperation, non¬compliance with medical treatment or unreliability.
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research/ Chicago Center for Facial Plastic Surgery
Locations (1):
- DeNova Research, Chicago, Illinois, United States

REFERENCES:
- See also: DeNova Research — http://www.denovaresearch.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcium Hydroxylapatite
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Blinded Evaluations of First Impression
Description: Upon completion of the study, 300 blinded evaluators will evaluate one of three binders comprised of a random visit photographs from baseline, optimal cosmetic result, and 1 month post optimal cosmetic result of 20 subjects. The 10-point (1=Not at all to 10=Extremely well) First Impression Scales consisting of 8 criteria. A score of 10 means favorable results and a score of 1 means unfavorable results.
Time Frame: After the 1-month post optimal correction visit for 20 subjects (averaged)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 19
score on a scale | 7.35 [6.15 to 8.50]

2. Primary Outcome: Self-esteem
Description: Self-esteem change will be determined by patient self-evaluation using the Heatherton & Polivy State Self-Esteem (HPSS). The primary variable will be measured as improvement in self-esteem from baseline self-evaluations.
  A 20-item scale that measures a participant's self-esteem at a given point in time. The 20 items are subdivided into 3 components of self-esteem: (1) performance self-esteem, social self-esteem, and appearance self-esteem. All items are answered using a 5-point scale (1= not at all, 2= a little bit, 3= somewhat, 4= very much, 5= extremely).
  Scores range from 20-100.
  Scores closer to 100 indicate a more favorable outcome.
Time Frame: 1 month
Population: All subjects completing indicated visit
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 19
units on a scale | 8.105 [7 to 9]

3. Primary Outcome: Self-esteem
Description: Self-esteem change will be determined by patient self-evaluation using the Heatherton & Polivy State Self-Esteem (HPSS). The primary variable will be measured as improvement in self-esteem from baseline self-evaluations.
  Self-esteem change will be determined by patient self-evaluation using the Heatherton & Polivy State Self-Esteem (HPSS). The primary variable will be measured as improvement in self-esteem from baseline self-evaluations.
  A 20-item scale that measures a participant's self-esteem at a given point in time. The 20 items are subdivided into 3 components of self-esteem: (1) performance self-esteem, social self-esteem, and appearance self-esteem. All items are answered using a 5-point scale (1= not at all, 2= a little bit, 3= somewhat, 4= very much, 5= extremely).
  Scores range from 20-100.
  Scores closer to 100 indicate a more favorable outcome.
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 19
score on a scale | 8.35 [7.55 to 9.35]

4. Secondary Outcome: Subject First Impression
Description: Each subject will complete a 10-point (1-Not at all to 10-Very Much) scale evaluating their own first impression at Baseline and 1-month post-OCR.
  First impression scores were recorded at baseline and 1-month post-OCR, and an average of the two scores were reported.
Time Frame: baseline and 1 month post-OCR (averaged)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 19
score on a scale | 7.35 [6.15 to 8.5]

5. Secondary Outcome: Assessment of Malar Deficiency
Description: Live subject malar deficiency severity will be rated by PI at Visits 1-4 according to the SOBER scale (Weeks 1-4 correspond to Visits 1-4).
  SOBER Scale (Solish Beer Remington Scale): is used to grade facial rhytids in the malar region.
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Extreme Grade 5: Extreme
  Scores closer to 1 is a more favorable outcome, while scores closer to 5 is a less favorable outcome
Time Frame: 1 month
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 19
score on a scale
  Visit 1 | 4.8 [4.1 to 5.0]
  Visit 2 | 4.2 [3.8 to 4.5]
  Visit 3 | 2.7 [2.3 to 3.1]
  Visit 4 | 1.6 [1.2 to 1.9]

6. Secondary Outcome: Aesthetic Improvement
Description: Investigator will complete GAIS (Global Aesthetic Improvement Scale) at Visits 2-4 comparing overall appearance of current visit's photo to baseline photo.
  Worse: -1 No Change: 0 Improved: 1 Much Improved: 2 Very Much Improved: 3
Time Frame: 1 month
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Calcium Hydroxylapatite
Number analyzed (Participants) | 19
score on a scale
  Visit 2 | 1.7 [1 to 3]
  Visit 3 | 1.9 [1 to 3]
  Visit 4 | 2.5 [1 to 3]

ADVERSE EVENTS:
Arm/Group | Calcium Hydroxylapatite
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No